CLINICAL TRIAL: NCT07066202
Title: Impact Assessment of SALSA (Sensing and Automation for Freedom, Security, Autonomy) Technological Solutions
Status: Recruiting | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Cascina Biblioteca Società Cooperativa Sociale (Unknown); Informatici Senza Frontiere APS (Unknown)
Responsible Party: Principal Investigator, Claudia Salatino, Bioengineer, Fondazione Don Carlo Gnocchi Onlus
Other Study IDs: CET 130/24, FDG 28_17/12/2024
Record Dates: First submitted 2025-02-17; First posted 2025-07-15 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Generalized Mental, Social and/or Motor Disability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention is planned in this study. Only the assessment of a specific condition. — No intervention is planned in this study. Only the assessment of a specific condition.

SUMMARY:
This study evaluates the impact of assistive technologies designed to improve the independence and safety of adults with disabilities living in shared residential environments. The project is called SALSA, which stands for "Sensorisation, Automation for Freedom, Security and Autonomy." It is being conducted in Milan, Italy, by a collaboration between Cascina Biblioteca Società Cooperativa Sociale, Fondazione Don Carlo Gnocchi ONLUS, and Informatici Senza Frontiere APS.

The goal of the study is to determine how well specific technologies-such as smart lighting systems and wearable monitoring devices-support residents' autonomy and daily functioning, while also reducing the workload for professional caregivers. These technologies are installed in apartments where people with mental, social, and/or physical disabilities live together with some support.

A total of 55 adults over the age of 18, all residents of Cascina Biblioteca's shared flats, will be enrolled. Technologies will be set up prior to the beginning of the trial. Data will be collected in three phases: before using the technologies (T0), after 30 days (T1), and after 60 days (T2). The evaluation includes personalized goals, physical environment metrics (like temperature, air quality, door use, and night movements), and ease of use of the systems by staff.

The study uses Goal Attainment Scaling (GAS) to track whether residents achieve their individual or group goals, and the System Usability Scale (SUS) to assess how user-friendly the technologies are from the caregivers' perspective. All data will be collected through structured webforms to reduce the chance of missing information and increase consistency. The study team will use both descriptive and inferential statistical methods to assess results over time.

A total of 55 adults over the age of 18, all residents of Cascina Biblioteca's shared flats, will be enrolled. Technologies will be set up prior to the beginning of the trial. Data will be collected in three phases: before using the technologies (T0), after 30 days (T1), and after 60 days (T2). The evaluation includes personalized goals, physical environment metrics (like temperature, air quality, door use, and night movements), and ease of use of the systems by staff.

The study uses Goal Attainment Scaling (GAS) to track whether residents achieve their individual or group goals, and the System Usability Scale (SUS) to assess how user-friendly the technologies are from the caregivers' perspective. All data will be collected through structured webforms to reduce the chance of missing information and increase consistency. The study team will use both descriptive and inferential statistical methods to assess results over time.

This research aims to provide practical insights into how technology can support adults with disabilities in more independent, safer living situations. It may also inform broader applications of these systems in similar care contexts. The protocol was approved by an Ethics Committee (CET 130/24; FDG 28_17/12/2024) and is in the data collection phase as of early 2025.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years of age;
* mental, social and/or motor disability;
* signature of consent for participation.

Exclusion Criteria:

* under 18 years of age;
* non-signature of consent to participation.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The impact assessment study will involve Cascina Biblioteca residents with the following characteristics: age over 18 and mental, social and/or motor disability.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Goal Attainment Scale (GAS) | Evaluations will be conducted at three time points: T0: Baseline (initial assessment) T1: 30 days after the baseline T2: 60 days after the baseline
  The Goal Attainment Scaling (GAS) is a scale used to measure how well individual therapy or intervention goals are achieved. It uses a 5-point scale ranging from -2 to +2, where each score reflects the degree to which the outcome met, exceeded, or fell short of expectations: +2: Outcome was much better than expected; +1: Outcome was somewhat better than expected; 0: Outcome was exactly as expected; -1: Outcome was somewhat below expectations; -2: Outcome was much worse than expected, possibly even below the starting point.
  This structured approach allows for personalized goal tracking and provides a standardized way to evaluate progress in a meaningful and quantifiable manner.

SECONDARY OUTCOMES:
Quantitative metrics | Evaluations will be conducted at three time points: T0: Baseline (initial assessment) T1: 30 days after the baseline T2: 60 days after the baseline
  In addition to the Goal Attainment Scaling (GAS), the study will collect a range of quantitative metrics to better understand the impact of innovative technological solutions on the daily lives of individuals with disabilities. These metrics will include environmental conditions (e.g., indoor temperature), safety-related indicators (e.g., number of emergency situations, unintended door openings, lack of ventilation), and the frequency of critical events (e.g., falls, water leaks). This data will provide objective context to complement the subjective assessment of goal achievement, allowing for a more comprehensive evaluation of the interventions' effectiveness and their influence on everyday living conditions.
System Usability Scale (SUS) | Evaluations will be conducted at three time points: T1: 30 days after the baseline T2: 60 days after the baseline
  The System Usability Scale (SUS) is a widely used tool for assessing user experience, specifically focusing on usability. It yields a score ranging from 0 to 100, where higher scores indicate a more favorable perception of usability. A SUS score above 68 is generally considered above average.
  How the SUS Score is Calculated:
  Collect Responses:
  Participants answer 10 items using a 5-point Likert scale (from 1 = strongly disagree to 5 = strongly agree).
  Score Odd-Numbered Items (1, 3, 5, 7, 9): subtract 1 from the participant's response.
  Score Even-Numbered Items (2, 4, 6, 8, 10): subtract the participant's response from 5.
  Sum the Adjusted Scores: add all the adjusted values together. Multiply by 2.5: the total is multiplied by 2.5 to obtain the final SUS score (ranging from 0 to 100).
  SUS Score Interpretation Guide: 0-50: Poor (Awful); 51-67: Below Average (Poor); 68-71: Marginal (Okay); 72-80: Good; 80 and above: Excellent.

CONTACTS AND LOCATIONS:
Locations (1):
- Cascina Biblioteca Società Cooperativa Sociale, Milan, Italy, Italy